CLINICAL TRIAL: NCT02408081
Title: Family-Focused Nursing for Elderly Medical Patients and Their Family: A Randomized Controlled Trial
Brief Title: Family Focused Nursing for Elderly Medical Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: not able to be completed
Sponsor: University of Southern Denmark (Other)
Collaborators: University Hospital, Gentofte, Copenhagen (Other)
Responsible Party: Principal Investigator, Birte Oestergaard, Associate professor, University of Southern Denmark
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: UNR-H-6-2014-109-5
Record Dates: First submitted 2015-03-31; First posted 2015-04-03 (Estimated); Last update posted 2017-10-27 (Actual); Status verified 2017-10

CONDITIONS: Depression
Keywords: Depression; Family functioning; Family Focused Nursing; Quality of life
MeSH Terms: conditions — Depression | interventions — Nursing; Aging

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment as usual (No Intervention): Pharmacological treatment, patient information and counselling according to international and national guidelines by health professionals specialized in elderly medical patients.
- Family Focused Nursing (Experimental): Family Focused Nursing and treatment as usual
  Interventions: Behavioral: Family Focused Nursing

INTERVENTIONS:
Behavioral: Family Focused Nursing — All patients receive treatment as usual. Additionally, patients in the intervention arm receives family focused nursing consultations which are structured as sessions focusing on change, improvement and/or maintenance of family function within cognitive, affective and behavioral knowledge. Each session is organized and individualized according to the wishes and needs for education and counseling of the families within a period of one months.
  Other Names: Family; Nursing; Elderly
  Arms: Family Focused Nursing

SUMMARY:
The purpose of this study is to determine whether Family Focused Nursing are effective in the treatment of elderly medical patients with respect to prevalence of depression

DETAILED DESCRIPTION:
Psychosocial issues such as lack of social support and symptoms of depression, are risk factors associated to readmission for elderly medical patients. Families with elderly members in general want to be involved in the caring and want to maintain a close relation to their elderly family member. However, disease in a single family can have a negative effect on all members and may result in dysfunction of the family. International guidelines recommend that the patient's relatives are involved in patient education as well as the treatment. Family interventions might contribute to decline depression and readmissions, besides enhanced quality of life and family function among elderly medical patients and their next of kin.

ELIGIBILITY:
Inclusion Criteria:

* acute hospitalized
* an expected hospitalization of minimum two days
* speak and understand Danish
* signed informed consent

Exclusion Criteria:

* dementia (evaluated by the Mini Mental State Examination [MMSE] < 24)
* terminally ill patients whose survival rate is assessed to be less than a month

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Change in depressive symptoms assessed by 9 points measured on the Geriatric Depression Scale | Baseline, 7 days and 6 months after the intervention
  The effect of intervention on primary outcome are investigated as longitudinal data at seven days and six month. The data are analysed using mixed models

SECONDARY OUTCOMES:
Change in family function score on Brief Family Assessment Measure III | 7 days and 6 months
  The effect of intervention on secondary outcome are investigated as longitudinal
Change in health related quality of life on Medical Outcomes Study Short Form, SF-8 | 7 days and 6 months
  The effect of intervention on secondary outcome are investigated as longitudinal
Change in time spent between hospitalization | 7 days and 6 months
  The effect of intervention on secondary outcome are investigated as longitudinal

CONTACTS AND LOCATIONS:
Overall Officials: Penille W Perboell, MHSc, Principal Investigator — University of Southern Denmark
Locations (1):
- University Hospital Gentofte, Copenhagen, Hellerup, Denmark

IPD SHARING:
Plan to Share IPD: Undecided